CLINICAL TRIAL: NCT03271450
Title: The Dabigatran, Apixaban, Rivaroxaban, Edoxaban, Warfarin Comparative Effectiveness Research Study
Brief Title: The DARE Warfarin CER Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Katsiaryna Bykov, PharmD, ScD, Instructor, Brigham and Women's Hospital
Other Study IDs: 2017P000215
Record Dates: First submitted 2017-08-24; First posted 2017-09-05 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Deep Venous Thrombosis; Pulmonary Embolism
Keywords: dabigatran; warfarin; apixaban; edoxaban; extended treatment; oral anticoagulant; rivaroxaban; comparative safety; comparative effectiveness
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (30):
- Continuer at 90 Days: Dabigatran
  Interventions: Drug: Dabigatran: extended treatment (e.g at least 90 days)
- Continuer at 180 Days: Dabigatran
  Interventions: Drug: Dabigatran: extended treatment (e.g at least 180 days)
- Continuer at 270 Days: Dabigatran
  Interventions: Drug: Dabigatran: extended treatment (e.g at least 270 days)
- Continuer at 90 Days: Apixaban
  Interventions: Drug: Apixaban: extended treatment (e.g at least 90 days)
- Continuer at 180 Days: Apixaban
  Interventions: Drug: Apixaban: extended treatment (e.g at least 180 days)
- Continuer at 270 Days: Apixaban
  Interventions: Drug: Apixaban: extended treatment (e.g at least 270 days)
- Continuer at 90 Days: Rivaroxaban
  Interventions: Drug: Rivaroxaban: extended treatment (e.g at least 90 days)
- Continuer at 180 Days: Rivaroxaban
  Interventions: Drug: Rivaroxaban: extended treatment (e.g at least 180 days)
- Continuer at 270 Days: Rivaroxaban
  Interventions: Drug: Rivaroxaban: extended treatment (e.g at least 270 days)
- Continuer at 90 Days: Edoxaban
  Interventions: Drug: Edoxaban: extended treatment (e.g at least 90 days)
- Continuer at 180 Days: Edoxaban
  Interventions: Drug: Edoxaban: extended treatment (e.g at least 180 days)
- Continuer at 270 Days: Edoxaban
  Interventions: Drug: Edoxaban: extended treatment (e.g at least 270 days)
- Continuer at 90 Days: Warfarin
  Interventions: Drug: Warfarin: extended treatment (e.g at least 90 days)
- Continuer at 180 Days: Warfarin
  Interventions: Drug: Warfarin: extended treatment (e.g at least 180 days)
- Continuer at 270 Days: Warfarin
  Interventions: Drug: Warfarin: extended treatment (e.g at least 270 days)
- Discontinuer at 90 Days: Dabigatran
  Interventions: Drug: Dabigatran: extended treatment (e.g at least 90 days)
- Discontinuer at 180 Days: Dabigatran
  Interventions: Drug: Dabigatran: extended treatment (e.g at least 180 days)
- Discontinuer at 270 Days: Dabigatran
  Interventions: Drug: Dabigatran: extended treatment (e.g at least 270 days)
- Discontinuer at 90 Days: Apixaban
  Interventions: Drug: Apixaban: extended treatment (e.g at least 90 days)
- Discontinuer at 180 Days: Apixaban
  Interventions: Drug: Apixaban: extended treatment (e.g at least 180 days)
- Discontinuer at 270 Days: Apixaban
  Interventions: Drug: Apixaban: extended treatment (e.g at least 270 days)
- Discontinuer at 90 Days: Rivaroxaban
  Interventions: Drug: Rivaroxaban: extended treatment (e.g at least 90 days)
- Discontinuer at 180 Days: Rivaroxaban
  Interventions: Drug: Rivaroxaban: extended treatment (e.g at least 180 days)
- Discontinuer at 270 Days: Rivaroxaban
  Interventions: Drug: Rivaroxaban: extended treatment (e.g at least 270 days)
- Discontinuer at 90 Days: Edoxaban
  Interventions: Drug: Edoxaban: extended treatment (e.g at least 90 days)
- Discontinuer at 180 Days: Edoxaban
  Interventions: Drug: Edoxaban: extended treatment (e.g at least 180 days)
- Discontinuer at 270 Days: Edoxaban
  Interventions: Drug: Edoxaban: extended treatment (e.g at least 270 days)
- Discontinuer at 90 Days: Warfarin
  Interventions: Drug: Warfarin: extended treatment (e.g at least 90 days)
- Discontinuer at 180 Days: Warfarin
  Interventions: Drug: Warfarin: extended treatment (e.g at least 180 days)
- Discontinuer at 270 Days: Warfarin
  Interventions: Drug: Warfarin: extended treatment (e.g at least 270 days)

INTERVENTIONS:
Drug: Dabigatran: extended treatment (e.g at least 90 days) — 90 days
  Groups: Continuer at 90 Days: Dabigatran; Discontinuer at 90 Days: Dabigatran
Drug: Dabigatran: extended treatment (e.g at least 180 days) — 180 days
  Groups: Continuer at 180 Days: Dabigatran; Discontinuer at 180 Days: Dabigatran
Drug: Dabigatran: extended treatment (e.g at least 270 days) — 270 days
  Groups: Continuer at 270 Days: Dabigatran; Discontinuer at 270 Days: Dabigatran
Drug: Apixaban: extended treatment (e.g at least 90 days) — 90 days
  Groups: Continuer at 90 Days: Apixaban; Discontinuer at 90 Days: Apixaban
Drug: Apixaban: extended treatment (e.g at least 180 days) — 180 days
  Groups: Continuer at 180 Days: Apixaban; Discontinuer at 180 Days: Apixaban
Drug: Apixaban: extended treatment (e.g at least 270 days) — 270 days
  Groups: Continuer at 270 Days: Apixaban; Discontinuer at 270 Days: Apixaban
Drug: Rivaroxaban: extended treatment (e.g at least 90 days) — 90 days
  Groups: Continuer at 90 Days: Rivaroxaban; Discontinuer at 90 Days: Rivaroxaban
Drug: Rivaroxaban: extended treatment (e.g at least 180 days) — 180 days
  Groups: Continuer at 180 Days: Rivaroxaban; Discontinuer at 180 Days: Rivaroxaban
Drug: Rivaroxaban: extended treatment (e.g at least 270 days) — 270 days
  Groups: Continuer at 270 Days: Rivaroxaban; Discontinuer at 270 Days: Rivaroxaban
Drug: Edoxaban: extended treatment (e.g at least 90 days) — 90 days
  Groups: Continuer at 90 Days: Edoxaban; Discontinuer at 90 Days: Edoxaban
Drug: Edoxaban: extended treatment (e.g at least 180 days) — 180 days
  Groups: Continuer at 180 Days: Edoxaban; Discontinuer at 180 Days: Edoxaban
Drug: Edoxaban: extended treatment (e.g at least 270 days) — 270 days
  Groups: Continuer at 270 Days: Edoxaban; Discontinuer at 270 Days: Edoxaban
Drug: Warfarin: extended treatment (e.g at least 90 days) — 90 days
  Groups: Continuer at 90 Days: Warfarin; Discontinuer at 90 Days: Warfarin
Drug: Warfarin: extended treatment (e.g at least 180 days) — 180 days
  Groups: Continuer at 180 Days: Warfarin; Discontinuer at 180 Days: Warfarin
Drug: Warfarin: extended treatment (e.g at least 270 days) — 270 days
  Groups: Continuer at 270 Days: Warfarin; Discontinuer at 270 Days: Warfarin

SUMMARY:
Approximately half a million Americans annually experience venous thromboembolic disease, including deep venous thrombosis (DVT) and pulmonary embolism (PE). Since 2010, four new oral anticoagulants have been approved for marketing in addition to the vitamin K antagonist warfarin. Very limited head-to-head data exists comparing these treatment options, leaving patients, clinicians, and other stakeholders with little guidance for selecting the best strategy that balances recurrence reduction with risk of bleeding. In the DARE Warfarin CER Study, the researchers compare all five currently available oral anticoagulant agents for the extended treatment of DVT and PE, as well as no extended treatment. This study also aims to evaluate whether treatment heterogeneity exists for specific populations, such as older patients or those with renal dysfunction. In a secondary aim, the study will also leverage a database of linked electronic health record-insurance claims to validate diagnosis definitions and account for potential residual confounding by factors unmeasured in claims data. As the patient population includes all Medicare novel anticoagulant users and large numbers of commercially insured and Medicaid patients, the results will likely be transportable to the majority of US patients experiencing a DVT or PE. Pursuant to the objectives of the Patient-Centered Outcomes Research Institute, a study advisory committee consisting of key stakeholders will be actively involved in the study design and dissemination of results.

ELIGIBILITY:
Inclusion criteria:

1. Inpatient stay with diagnosis code of DVT/PE (see Appendix A), 1/1/2010 - 9/30/2015 for which the patient has at least 365 days continuous medical and pharmacy eligibility prior and no other inpatient stays with DVT/PE diagnosis. Set discharge date as index diagnosis date. Take only the first eligible episode for a patient, if multiple.
2. Prescription fill for an anticoagulant [generic name=dabigatran (150mg), apixaban (2.5mg, 5mg, 10mg), rivaroxaban (15mg, 20mg), edoxaban (30mg, 60mg), or warfarin] within 30 days of and including index diagnosis date. Set earliest anticoagulant prescription as index generic and date as index rx date.
3. No anticoagulant prescription fill in the 365 days prior to index diagnosis date.
4. Continuous enrollment and use of an anticoagulant for the first 90 days including and following the index rx date, defined as no gaps in therapy >7 days. For each patient, assign a variable to indicate whether the patient filled an anticoagulant with a different generic name as index during this period.

Exclusion Criteria:

1. Any safety outcome between index diagnosis date and index rx date + 90, defined as: intracranial bleed, gastrointestinal bleed, or other major bleed.
2. Any DVT/PE between index diagnosis date and index rx date + 90.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort derived from a commercial database, MarketScan, and Medicare Research Identifiable Files using data from 2009-2015. Cohort data will be updated as new data come in through 2019.
Sampling Method: Non-Probability Sample
Enrollment: 416000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Composite Safety Outcome: Intracranial bleed, Gastrointestinal bleed, Other Major bleed | 1-2 Years
  Defined as a new episode of either Intracranial bleed, Gastrointestinal bleed or another Major bleed event during follow-up.
Composite Effectiveness Outcome: Deep Venous Thrombosis, Pulmonary Embolism | 1-2 Years
  Defined as a new episode of either Deep Venous Thrombosis or Pulmonary Embolism during follow-up.
Death | 1-2 Years
  Measured after index prescription date + 90 days and on date on which the event occurred and defined as hospitalization with discharge status code of: 20, 22-29, 40-42
Composite safety and effectiveness outcome | 1-2 years
  defined as earlier of safety or DVT/PE outcomes
Composite safety and effectiveness outcome, including death | 1-2 years
  Measured after index prescription date + 90 days and on date on which the event occurred and defined as hospitalization with discharge status code of: 20, 22-29, 40-42

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krumme AA, Pawar A, Schneeweiss S, Glynn RJ, Choudhry NK, Kulldorff M, Ortiz AS, Avorn J, Gagne JJ. Study protocol for the dabigatran, apixaban, rivaroxaban, edoxaban, warfarin comparative effectiveness research study. J Comp Eff Res. 2018 Jan;7(1):57-66. doi: 10.2217/cer-2017-0053. Epub 2017 Dec 21. PMID 29264930